CLINICAL TRIAL: NCT01318694
Title: A Randomized, Double-blind, Placebo-controlled Trial of the Efficacy and Safety of DEB025/Alisporivir in Combination With Peg-IFNα2a and Ribavirin in Hepatitis C Genotype 1 Treatment-naïve Patients
Brief Title: Efficacy and Safety of Alisporivir Triple Therapy in Chronic Hepatitis C Genotype 1 Treatment-naïve Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDEB025A2301; 2010-022867-37 (EudraCT Number)
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Results first posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis C
Keywords: Chronic hepatitis C; Cyclophilin inhibitor
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — alisporivir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Treatment Arm A (Experimental): Alisporivir (ALV) 600 mg twice daily (BID) with Peginterferon alfa-2a (PEG) and ribavirin (RBV) for 1 week, followed by an additional 23 or 47 weeks according to response-guided treatment duration (RGT):
  * Participants with a viral load below the level of detection (< LOD) at Week 4 stop study treatment after 24 weeks
  * Participants with a viral load ≥ LOD at Week 4 complete 48 weeks of study treatment
  Interventions: Drug: Alisporivir; Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Treatment Arm B (Experimental): Alisporivir (ALV) 400 mg twice daily (BID) with PEG and RBV for 24 or 48 weeks according to response-guided treatment duration (RGT)
  Interventions: Drug: Alisporivir; Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Treatment Arm C (Experimental): Alisporivir (ALV) 600 mg BID with PEG and RBV for 1 week, followed by 600 mg once daily (QD) for 47 weeks
  Interventions: Drug: Alisporivir; Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Treatment Arm D (Active Comparator): ALV Placebo with PEG and RBV for 48 weeks
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin; Drug: ALV Placebo

INTERVENTIONS:
Drug: Alisporivir — ALV 200 mg soft gel capsules administered orally
  Other Names: DEB025; ALV
  Arms: Treatment Arm A; Treatment Arm B; Treatment Arm C
Drug: Peginterferon alfa-2a — PEG 180 μg administered via subcutaneous (s.c.) injection once weekly
  Other Names: Pegasys®; PEG
Drug: Ribavirin — RBV 200 mg tablets (weight-based dose: < 75 mg = 1000 mg/day; ≥ 75 kg = 1200 mg/day) administered orally in a divided daily dose
  Other Names: Copegus®; RBV
Drug: ALV Placebo — ALV placebo soft gel capsules administered orally
  Other Names: Placebo
  Arms: Treatment Arm D

SUMMARY:
This study will assess the safety and efficacy of alisporivir (ALV; DEB025) triple therapy [i.e., when added to peginterferon alfa-2a (PEG) and ribavirin (RBV)] to optimize treatment in treatment-naïve participants with hepatitis C virus (HCV) genotype 1 (GT1)

ELIGIBILITY:
Inclusion criteria:

* Chronic HCV infection
* HCV genotype 1
* No previous treatment for hepatitis C infection
* Serum HCV RNA level ≥ 1000 IU/ml assessed by quantitative polymerase chain reaction or equivalent at screening, no upper limit
* Liver evaluation prior to baseline: liver biopsy within 3 years or Fibroscan within 6 months

Exclusion criteria:

* HCV genotype different from genotype 1 or co-infection with other HCV genotype
* Co-infection with Hepatitis B or HIV
* Any other cause of relevant liver disease other than HCV
* Presence or history of hepatic decompensation
* Alanine aminotransferase (ALT) ≥ 10 times upper limit of normal (ULN), more than 1 episode of elevated bilirubin (> ULN) in past 6 months

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1081 (Actual)
Dates: Start 2011-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (120):
- United States (26):
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Oakland, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Ventura, California
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Maitland, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Shreveport, Louisiana
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Newark, New Jersey
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Fayetteville, North Carolina
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Fairfax, Virginia
  - Novartis Investigative Site, Newport News, Virginia
- Argentina (3):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
- Australia (6):
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Kingswood, New South Wales
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Greenslopes, Queensland
  - Novartis Investigative Site, Fitzroy, Victoria
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
- Canada (5):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Downsview, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
- France (5):
  - Novartis Investigative Site, Clichy
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (10):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
- Novartis Investigative Site, Hong Kong, Hong Kong, Hong Kong
- Hungary (6):
  - Novartis Investigative Site, Békéscsaba
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Székesfehérvár
- Italy (11):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Napoli
- Mexico (2):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
- Poland (5):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Chorzów
  - Novartis Investigative Site, Kielce
  - Novartis Investigative Site, Lódz
- Novartis Investigative Site, San Juan, Puerto Rico
- Romania (7):
  - Novartis Investigative Site, Bucharest, District 1
  - Novartis Investigative Site, Bucharest, District 3
  - Novartis Investigative Site, Iași, Iaşi
  - Novartis Investigative Site, Iași, Jud. Iasi
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Craiova
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- South Korea (7):
  - Novartis Investigative Site, Busan, Busan
  - Novartis Investigative Site, Yangsan, Gyeongsangnam-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Kyunggi, Kyeonggi
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Pusan
- Spain (5):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Valencia, Valencia
- Taiwan (6):
  - Novartis Investigative Site, Chiayi City, Taiwan
  - Novartis Investigative Site, Niaosong Township, Taiwan
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Douliu
  - Novartis Investigative Site, Kaohsiung City
- Thailand (4):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Khon Kaen
  - Novartis Investigative Site, Songkhla
- United Kingdom (4):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Nottingham
- Vietnam (2):
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 1580 patients screened at multiple global sites, 1081 (68.4%) were randomized and 499 (31.6%) discontinued from the study prior to randomization.
Pre-assignment Details: Due to mis-randomization, four patients did not have a baseline visit and never started study medications. They were included in screened and randomized, but excluded from the Full Analysis Set and the Safety Set.
Groups:
- Treatment Arm A: Alisporivir (ALV) 600 mg twice daily (BID) with Peginterferon alfa-2a (PEG) and ribavirin (RBV) for 1 week, followed by an additional 23 or 47 weeks according to response-guided treatment duration (RGT)
Period: Overall Study
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D
Started | 275 | 270 | 268 | 268
Full Analysis Set | 274 | 270 | 265 | 268
Safety Set | 273 | 268 | 265 | 265
Completed | 223 | 212 | 225 | 200
Not Completed | 52 | 58 | 43 | 68

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS), defined as all participants to whom study treatment was correctly assigned.
Groups:
- Treatment Arm A: Alisporivir (ALV) 600 mg BID with PEG and RBV for 1 week, followed by an additional 23 or 47 weeks according to RGT
- Treatment Arm B: Alisporivir (ALV) 400 mg BID with PEG and RBV for 24 or 48 weeks according to RGT
- Treatment Arm C: Alisporivir (ALV) 600 mg BID with PEG and RBV for 1 week, followed by 600 mg QD for 47 weeks
- Total: Total of all reporting groups
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D | Total
Number analyzed (Participants) | 274 | 270 | 265 | 268 | 1077
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (11.08) | 45.8 (11.95) | 45.5 (12.15) | 46.3 (11.53) | 45.9 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 106 | 134 | 114 | 467
  Male | 161 | 164 | 131 | 154 | 610

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Sustained Virologic Response (SVR) 12 Weeks After the End of Treatment (SVR12)
Description: SVR12 was defined as hepatitis C virus (HCV) RNA laboratory value below the level of quantification (< LOQ; i.e., 25 IU/ml) 12 weeks after the end of treatment.
Time Frame: 12 weeks after the end of treatment
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D
Number analyzed (Participants) | 274 | 270 | 265 | 268
percentage of participants | 68.6 | 68.9 | 69.4 | 52.5

2. Secondary Outcome: Percentage of Participants Who Achieved SVR 24 Weeks After the End of Treatment (SVR24)
Description: SVR24 was defined as HCV RNA laboratory value < LOQ 24 weeks after the end of treatment.
Time Frame: 24 weeks after the end of treatment
Population: Participants in the Full Analysis Set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D
Number analyzed (Participants) | 273 | 268 | 265 | 265
percentage of participants | 68.5 | 69.0 | 68.3 | 51.7

3. Secondary Outcome: Percentage of Participants With Rapid Virologic Response (RVR) After 4 Weeks of Treatment (RVR4)
Description: RVR4 was defined as serum HCV RNA < LOQ after 4 weeks of treatment.
Time Frame: after 4 weeks of treatment
Population: Participants in the Full Analysis Set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D
Number analyzed (Participants) | 268 | 258 | 258 | 261
percentage of participants | 60.1 | 72.5 | 56.6 | 28.4

4. Secondary Outcome: Percentage of Participants With Early Virologic Response (EVR) After 12 Weeks of Treatment
Description: EVR was defined as a ≥ 2 log10 decrease in HCV RNA or HCV RNA < LOQ after 12 weeks of treatment.
Time Frame: after 12 weeks of treatment
Population: Participants in the Full Analysis Set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D
Number analyzed (Participants) | 259 | 242 | 247 | 256
percentage of participants | 97.7 | 98.3 | 99.6 | 89.8

5. Secondary Outcome: Percentage of Participants With Partial Early Virologic Response (pEVR) After 12 Weeks of Treatment
Description: pEVR was defined as a ≥ 2 log10 decrease in HCV RNA and still detectable (≥ LOQ) after 12 weeks of treatment.
Time Frame: after 12 weeks of treatment
Population: Participants in the Full Analysis Set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D
Number analyzed (Participants) | 259 | 242 | 247 | 256
percentage of participants | 8.1 | 2.1 | 10.5 | 19.5

6. Secondary Outcome: Percentage of Participants With Complete Early Virologic Response (cEVR) After 12 Weeks of Treatment
Description: cEVR was defined as serum HCV RNA < LOQ after 12 weeks of treatment.
Time Frame: after 12 weeks of treatment
Population: Participants in the Full Analysis Set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D
Number analyzed (Participants) | 259 | 242 | 247 | 256
percentage of participants | 89.6 | 96.3 | 89.1 | 70.3

7. Secondary Outcome: Percentage of Participants With Extended Rapid Virologic Response (eRVR) From 4 to 12 Weeks of Treatment
Description: eRVR was defined as achieving RVR4 and maintaining HCV RNA < LOQ until Week 12.
Time Frame: from 4 to 12 weeks of treatment
Population: Participants in the Full Analysis Set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D
Number analyzed (Participants) | 259 | 242 | 247 | 256
percentage of participants | 60.2 | 71.1 | 56.7 | 28.1

8. Secondary Outcome: Percentage of Participants With End of Treatment Response (ETR) at Treatment End Within 48 Weeks
Description: ETR was defined as serum HCV RNA < LOQ at treatment end (completed or prematurely discontinued).
Time Frame: at treatment end within 48 weeks
Population: Participants in the Full Analysis Set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D
Number analyzed (Participants) | 271 | 268 | 264 | 265
percentage of participants | 88.2 | 87.7 | 87.5 | 80.0

9. Secondary Outcome: Percentage of Participants With Alanine Aminotransferase (ALT) Abnormalities Within 48 Weeks
Description: ALT abnormalities were summarized as participants who had either:
  * ALT > 2 x upper limit of normal (ULN) during the study and > 2 x ULN at baseline
  * ALT > 3 x ULN during the study and > 2 x ULN at baseline
Time Frame: within 48 weeks
Population: Participants in the Safety Set, defined as having received at least one dose of study medication, with available data
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D
Number analyzed (Participants) | 271 | 267 | 264 | 264
percentage of participants
  > 2 x ULN and > 2 x baseline | 1.5 | 0.4 | 1.9 | 1.5
  > 3 x ULN and > 2 x baseline | 0.7 | 0.0 | 1.5 | 0.8

10. Secondary Outcome: Percentage of Participants With Grade 3 or 4 Anemia During Treatment Within 48 Weeks
Description: Grading was according to the Modified Division of Microbiology & Infectious Diseases (DMID) Toxicity Tables (version 2.0).
  Participants with multiple abnormalities were counted only once in the worst category.
Time Frame: within 48 weeks
Population: Participants in the Safety Set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D
Number analyzed (Participants) | 271 | 267 | 264 | 264
percentage of participants
  Grade 3 | 1.8 | 3.4 | 0.8 | 1.9
  Grade 4 | 0.0 | 0.4 | 0.0 | 0.0

11. Secondary Outcome: Percentage of Participants With Grade 3 or 4 Neutropenia During Treatment Within 48 Weeks
Description: Grading was according to the DMID Toxicity Tables (version 2.0). Participants with multiple abnormalities were counted only once in the worst category.
Time Frame: within 48 weeks
Population: Participants in the Safety Set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D
Number analyzed (Participants) | 270 | 263 | 264 | 264
percentage of participants
  Grade 3 | 24.4 | 24.7 | 23.1 | 12.9
  Grade 4 | 4.4 | 8.0 | 7.2 | 2.7

12. Secondary Outcome: Percentage of Participants With Grade 3 or 4 Thrombocytopenia During Treatment Within 48 Weeks
Description: as for outcome 11
Time Frame: within 48 weeks
Population: Participants in the Safety Set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D
Number analyzed (Participants) | 270 | 265 | 264 | 264
percentage of participants
  Grade 3 | 6.7 | 21.9 | 12.5 | 1.9
  Grade 4 | 0.0 | 1.1 | 0.0 | 0.0

ADVERSE EVENTS:
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Treatment Arm D
Serious Adverse Events (participants affected / at risk) | 24/273 | 28/268 | 21/265 | 28/265
Other Adverse Events (participants affected / at risk) | 256/273 | 261/268 | 250/265 | 242/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm A (N=273) | Treatment Arm B (N=268) | Treatment Arm C (N=265) | Treatment Arm D (N=265)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 2 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Dacryoadenitis acquired (Eye disorders) | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 3 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 0
Drug interaction (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Lipogranuloma (General disorders) | 1 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 1 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Cervicitis (Infections and infestations) | 0 | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Nasal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Salpingo-oophoritis (Infections and infestations) | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1
Mania (Psychiatric disorders) | 0 | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
Bartholinitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 3 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm A (N=273) | Treatment Arm B (N=268) | Treatment Arm C (N=265) | Treatment Arm D (N=265)
Anaemia (Blood and lymphatic system disorders) | 113 | 124 | 91 | 88
Leukopenia (Blood and lymphatic system disorders) | 48 | 27 | 48 | 27
Lymphopenia (Blood and lymphatic system disorders) | 15 | 7 | 16 | 8
Neutropenia (Blood and lymphatic system disorders) | 86 | 80 | 86 | 67
Thrombocytopenia (Blood and lymphatic system disorders) | 47 | 73 | 49 | 16
Hypothyroidism (Endocrine disorders) | 17 | 22 | 23 | 12
Ocular icterus (Eye disorders) | 11 | 14 | 5 | 4
Abdominal pain upper (Gastrointestinal disorders) | 18 | 24 | 22 | 15
Constipation (Gastrointestinal disorders) | 12 | 17 | 7 | 12
Diarrhoea (Gastrointestinal disorders) | 30 | 27 | 38 | 37
Dyspepsia (Gastrointestinal disorders) | 23 | 17 | 32 | 18
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 | 9 | 7 | 15
Nausea (Gastrointestinal disorders) | 66 | 67 | 62 | 45
Vomiting (Gastrointestinal disorders) | 26 | 39 | 29 | 19
Asthenia (General disorders) | 43 | 46 | 46 | 48
Chills (General disorders) | 23 | 30 | 33 | 21
Fatigue (General disorders) | 84 | 99 | 87 | 86
Influenza like illness (General disorders) | 56 | 52 | 38 | 40
Injection site erythema (General disorders) | 14 | 10 | 17 | 8
Irritability (General disorders) | 19 | 16 | 21 | 22
Pyrexia (General disorders) | 78 | 93 | 82 | 74
Hyperbilirubinaemia (Hepatobiliary disorders) | 32 | 61 | 25 | 2
Jaundice (Hepatobiliary disorders) | 7 | 20 | 3 | 1
Nasopharyngitis (Infections and infestations) | 9 | 9 | 17 | 12
Upper respiratory tract infection (Infections and infestations) | 16 | 5 | 16 | 13
Urinary tract infection (Infections and infestations) | 11 | 14 | 11 | 8
Weight decreased (Investigations) | 24 | 28 | 26 | 18
Decreased appetite (Metabolism and nutrition disorders) | 61 | 59 | 58 | 42
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 11 | 23 | 22 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 | 35 | 39 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 14 | 15 | 20
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 17 | 7 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 59 | 53 | 56 | 52
Dizziness (Nervous system disorders) | 33 | 34 | 25 | 30
Dysgeusia (Nervous system disorders) | 14 | 22 | 13 | 11
Headache (Nervous system disorders) | 91 | 94 | 94 | 80
Anxiety (Psychiatric disorders) | 17 | 20 | 25 | 29
Depression (Psychiatric disorders) | 20 | 29 | 28 | 23
Insomnia (Psychiatric disorders) | 49 | 61 | 50 | 60
Cough (Respiratory, thoracic and mediastinal disorders) | 47 | 54 | 59 | 53
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 37 | 26 | 23 | 26
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 25 | 15 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 13 | 19 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 60 | 45 | 57 | 47
Dry skin (Skin and subcutaneous tissue disorders) | 21 | 23 | 31 | 22
Pruritus (Skin and subcutaneous tissue disorders) | 58 | 55 | 49 | 54
Rash (Skin and subcutaneous tissue disorders) | 46 | 40 | 45 | 45
Hypertension (Vascular disorders) | 31 | 50 | 34 | 7

LIMITATIONS AND CAVEATS:
In April 2012, ALV and placebo were discontinued in all participants. Participants remained on PEG and RBV treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other